### **J-SUPREME II Clinical Trial**

A Prospective, Multicenter, Single-arm Clinical Trial of JetStream Atherectomy System for the Treatment of Japanese Patients with Symptomatic OcclUsive Atherosclerotic Lesions in the SuPeRficial FEmoral and/ or ProxiMal PoplitEal Arteries

### CLINICAL INVESTIGATION PLAN

S2450

### **Sponsored By**

Boston Scientific Japan K.K. 4-10-2, Nakano Nakano-ku Tokyo 164-0001, Japan

*This protocol contains confidential information* for use by the Investigators and their designated representatives participating in this clinical investigation. The protocol should be held confidential and maintained in a secure location.

Do not copy or distribute without written permission from Boston Scientific Corporation.

### **Contact Information**

| Role | Contact |
|---|---|
| Investigational Centers | A list of investigational sites is maintained and provided as a separate attachment to the protocol. |
| Vendors/Labs | A list of vendors/laboratories involved in the trial is maintained by the sponsor and will be provided to investigational sites. |

Original Release: January 29, 2019

Current Version: July 4, 2019

| | | N/A | |
|---|---|---|---|
| CIUZ 14 AUDICIO I CIUNIO CIUN A 17 ZIUN CIUN A 17 ZIUN CIUN A 17 ZIUN CIUN CIUN CIUN CIUN CIUN CIUN CIUN C | | | |
| | Revision Protocol Date Version | | July 4, 2019 |
| | Revision<br>Version | | Э |

## 2. Protocol Synopsis

| J-SUPREME II: A Pro<br>System for the Treatm<br>Lesions in the Superfic | ent of Japane | se Patients with Sympto | omatic Occl | usive Atheroscle | |
|---|---|---|---|---|---|
| Study Objective(s) | Atherectomy symptomatic | he safety and effectivene<br>System (Jetstream) for<br>occlusive atherosclero<br>and/ or proximal poplite | the treatm | ent of Japanese p<br>in native superfic | atients with |
| Test Device and device Sizes | 1 | n® Atherectomy System:<br>ctive removal of atheros | • | | |
| | Jetstream At | herectomy System | | | |
| | 1. Jetstream Model | Catheter Tip Diameter | Catheter<br>Length | Min.Introducer<br>Size | Max.<br>Guidewire<br>Diameter |
| | SC 1.6 | 1.6 mm | 145 cm | 7 Fr | |
| | SC 1.85 | 1.85 mm | 145 cm | 7 F1 | 0.014 inch |
| | XC 2.1/3.0 | 2.1 mm (Blade Down)<br>3.0 mm (Blade Up) | 135 cm | 7 Fr | 0.014 men |
| | XC 2.4/3.4 | 2.4 mm (Blade Down)<br>3.4 mm (Blade Up) | 120 cm | | |
| | 2. Jetstream | Console | | | |
| <b>Control Device</b> | NA | | | | |
| Study Design | the Jetstream atherosclerot | e, multicenter, single-arm<br>Atherectomy System is<br>ic lesions ≤150 mm in lea<br>ith symptoms classified | n the treatm | ent of symptomat in the femoropopl | cic occlusive |
| Planned Number of<br>Subjects | Thirty-one (31) subjects will be enrolled. | | | | |
| Planned Number of<br>Investigational Sites/<br>Countries | Up to 4 investigational sites in Japan may enroll subjects. | | | | |
| Primary Endpoint | Lesion succe | effective endpoint is the ess is defined as the case | | | x procedure. |
| | After dilatati | on with DCB: | | | |



| Follow-up Schedule | <ul> <li>Subjects will be evaluated at 1 and 6 months post-index procedure.</li> <li>Subjects who are enrolled but the Jetstream Atherectomy System is not used will be followed through the 1-month follow-up visit only.</li> <li>Assessment of the primary endpoint will occur at the index procedure.</li> <li>All follow-up visits will be conducted in the office/clinic.</li> <li>Planned protocol-required testing includes the following:</li> <li>Angiography during the index procedure to assess procedural success and occurrence of emboli.</li> <li>IVUS during the index procedure to assess lesion</li> <li>DUS at the 1-month and 6-months follow-up visits to assess lesion and vessel patency</li> </ul> |
|---|---|
| Study Duration | The trial will be considered complete (with regards to the primary endpoint) after all enrolled subjects have completed the index procedure, are discontinued prior to completion of the procedure or have died. The trial will be considered complete (with regards to all follow-up) after all enrolled subjects have completed the 6 month follow-up visit, are discontinued prior to 6 month follow-up visit, have died, or the last 6 month follow-up visit window is closed. It is estimated that it will take approximately 1 year to complete this trial. |
| Key Inclusion<br>Criteria | <ol> <li>≥20 years of age</li> <li>An acceptable candidate for percutaneous intervention and/or emergency surgery.</li> <li>Willing and able to provide consent before any study specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits</li> <li>Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3 or 4</li> <li>Stenotic, restenotic or occlusive lesion(s) located in the native SFA and/or PPA of which meet all of the following criteria*: <ol> <li>Severely calcified lesions with degree of stenosis ≥70% by visual angiographic assessment</li> </ol> </li> <li>c. Guidewire must cross lesion(s) within the true lumen, without a subintimal course by physician's discretion based on visual estimate</li> <li>d. Vessel diameter ≥3.0 mm and ≤6.0 mm by visual estimate</li> <li>e. Total lesion length (or series of lesions) ≤150 mm by visual estimate</li> <li>f. Target lesion located at least 3 cm above the inferior edge of the femur by visual estimate</li> </ol> |

| | 1 age 7 01 30 |
|---|---|
| | 6. Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis by visual estimate) to the ankle or foot with no planned intervention |
| Key Exclusion<br>Criteria | 1. Target lesion must be one and decided by physician's discretion in the case that eligible lesions exist in both limbs |
| | 2. Target lesion/vessel with in-stent restenosis |
| | 3. Target lesion/vessel previously treated with any stent placement prior to the procedure |
| | 4. Use of atherectomy, laser or other debulking devices other than the Jetstream System, CTO devices or cutting balloon, Angioscore or similar devices, or ultra-high pressure balloon in the target limb SFA/PPA during the index procedure |
| | 5. History of major amputation in the target limb |
| | 6. Life expectancy less than 12 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the clinical trial, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the clinical trial |
| | 7. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated |
| | 8. Known hypersensitivity/allergy to the investigational atherectomy system or protocol related therapies (e.g., nitinol, stainless steel or other stent materials, and antiplatelet or anticoagulant, thrombolytic medications) |
| | 9. Subject has a history of coagulopathy or hypercoagulable bleeding disorder |
| | 10 Subject with untreatable hemorrhagic disease or platelet count <80,000 mm <sup>3</sup> or >600,000 mm <sup>3</sup> as baseline assessment. |
| | 11. Being on peritoneal dialysis |
| | 12. History of myocardial infarction, or stroke/cerebrovascular accident (CVA) within 6 months prior to study enrollment |
| | 13. Unstable angina pectoris at the time of the enrollment |
| | 14. Pregnancy and/or breast feeding |
| | 15. Current participation in another investigational drug or device clinical study that has not completed the primary endpoint at the time of enrollment or that clinically interferes with the current study endpoints (Note: studies requiring extended follow-up for products that were investigational, but have become commercially available since then are not considered investigational studies.) |
| | 16. Septicemia at the time of enrollment |
| | 17. Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure |
| | 18. Presence of aneurysm in the target vessel |
| | 19. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to the index procedure |



### 3. Table of Contents

| 1. | Title | Page | 1 |
|-----|-------|--------------------------------------------------|----|
| 2. | Proto | ocol Synopsis | 4 |
| 3. | Table | e of Contents | 9 |
| | 3.1. | Table of Figures | 11 |
| | 3.2. | Table of Tables | 11 |
| 4. | Intro | duction | 13 |
| | 4.1. | Background of development | 13 |
| | 4.2. | Clinical Study Summary | 13 |
| | | 4.2.1. Summary of Pathway PVD clinical trial | 13 |
| | | 4.2.2. Summary of J-SUPREME clinical trial | |
| 5. | Devi | ce Description | 15 |
| | 5.1. | Jetstream Atherectomy Catheter | 16 |
| | 5.2. | Jetstream Console | 17 |
| | 5.3. | Device Labeling of investigational device | 17 |
| 6. | Stud | y Objectives and Endpoints | 17 |
| | 6.1. | Study Objective | 17 |
| | 6.2. | Primary Endpoint | 17 |
| | 6.3. | Additional Endpoint | 18 |
| 7. | Stud | y Design | 18 |
| | 7.1. | Scale and Duration | 18 |
| 8. | Subje | ect Selection | 20 |
| • | 8.1. | Study Population and Eligibility | |
| | 8.2. | Inclusion Criteria | |
| | 8.3. | Exclusion Criteria | |
| 9. | | ect Accountability | |
| | 9.1. | Point of Enrollment | |
| | 9.2. | Withdrawal | |
| | 9.3. | Lost to Follow-Up | |
| | 9.4. | End-of- Study Definition | |
| 10. | Study | y Methods | |
| | 10.2. | Study Candidate Screening | 25 |
| | | 10.2.1. Strategies for Recruitment and Retention | |
| | 10.3. | Informed Consent | 25 |

| | 10.13 | .Follow-up | 28 |
|---|---|---|---|
| 11. | Statis | stical Considerations | . 29 |
| | 11.1. | Endpoints | 29 |
| | 11.2. | General Statistical Methods | 30 |
| | | 11.2.1. Analysis Sets | 30 |
| | | 11.2.2. Control of Systematic Error/Bias | 30 |
| | | 11.3.2. Interim Analyses | 31 |
| | | AA O A hostification of Dealing | 0.4 |
| | | 11.3.4. Justification of Pooling | .31 |
| | | 11.3.6. Other Analyses | 20 |
| | | 11.3.7. Changes to Planned Analyses | |
| 12 | Data | Management | |
| 12. | | Data Collection, Processing, and Review | 32 |
| | | Data Retention | |
| | | Core Laboratories | |
| 12 | | | |
| | | ations | |
| | | e/Equipment Accountability | |
| 15. | _ | oliance | |
| | 15.1. | Statement of Compliance | 34 |
| | 15.2. | Investigator Responsibilities | |
| | | 15.2.1. Delegation of Responsibility | |
| | | Institutional Review Board | |
| | 15.4. | Sponsor Responsibilities | |
| | | 15.4.1. Role of Boston Scientific Japan K.K. Representatives | |
| | | Reimbursement and Compensation | |
| 16. | Monit | toring | . 37 |

| | | | Ļ |
|---|---|---|---|
| | 172 | Risks associated with Participation in the Clinical Study | 38 |
| | | Possible Interactions with Concomitant Medical Treatments | |
| | | Risk Minimization Actions | |
| | | Anticipated Benefits | |
| | | Risk to Benefit Rationale | |
| 18. | Safety | Reporting | 39 |
| | 18.1. I | Reportable Events by investigational site to Boston Scientific | 39 |
| | 18.5. I | Boston Scientific Device Deficiencies | 44 |
| | 18.6. I | Reporting to Regulatory Authorities / IRBs / Investigators | 44 |
| 19. | Inform | ed Consent | 45 |
| 20. | Comm | ittees | 46 |
| | 20.1. I | Executive Committee | 46 |
| 0.4 | | | 4.5 |
| 21. | - | nsion or Termination | |
| | | Premature Termination of the Study | |
| | | 21.1.1. Criteria for Premature Termination of the Study | |
| | | Requirements for Documentation and Subject Follow-up | |
| | | Criteria for Suspending/Terminating a Study Site | |
| 22. | | ation Policy | |
| 24. | Abbre | viations and Definitions | 49 |
| | 24.1. | Abbreviations | 49 |
| 3.1. | Tak | ole of Figures | |
| Fiaı | ıre 5-1∶ | Jetstream Atherectomy System | 16 |
| _ | | Jetstream Catheter Tip | |
| 3.2. | | ble of Tables | |
| | | Jetstream Specifications | |
| Tab | le 8-1: | Inclusion Criteria | 20 |

### 4. Introduction

### 4.1. Background of development

Peripheral arterial disease (PAD) is a chronic arterial occlusive disease of the lower extremities caused by arteriosclerosis. The most common clinical symptom of PAD is intermittent claudication, and as the disease progresses, serious problems such as physical disability and significant deterioration of quality of life (QOL) can develop. For these PAD patients, various therapies have been tried including medication, exercise therapy, endvascular therapy (EVT) and surgical revascularization. With regards to the therapies for PAD, especially, femoropopoliteal artery, EVT has been one of the treatment options and treatment with balloon or stent is common in Japan. Since Drug-coated balloon (DCB) was approved in Japan in August, 2017,



Jetstream Atherectomy System was approved under 510(K) for the Pathway PV System, a first-generation model, in July 2008, and later in April 2013, for the current model. Jetstream Atherectomy System was also granted a CE mark in September 2013 and is currently marketed in the United States, Europe, Canada, Australia, and other regions.

### 4.2. Clinical Study Summary

#### 4.2.1. Summary of Pathway PVD clinical trial

The pathway PVD clinical study was a prospective, multicenter, single arm study conducted using the Pathway PV System, a first-generation model of Jetstream, in which a total of 172 subjects were enrolled at 9 investigational sites in Germany, Austria, and Belgium.

The primary safety endpoints of this study was the free rate for serious adverse device effects (SADEs) and target lesion revascularization (TLR) in the 6-month post-procedure period. The primary efficacy endpoint was the procedural success rate (defined as reduction in lesion stenosis, that is, the difference between the stenosis diameter prior to treatment with Jetstream and the stenosis diameter following treatment with Jetstream [absolute mean percentage]). Target lesions had reference vessel diameters ranging from 3–5 mm (visual estimation), total lesion lengths (alone or series of lesions) up to 10 cm for the superficial femoral and popliteal arteries as well as up to 3 cm for the tibial and fibular arteries (the superficial femoral artery), and lesions in the infrapopliteal and popliteal artery (Rutherford categories 1–5 or equivalent).

The free rate for SADEs and TLR for the 6-month post-procedure period, the primary safety endpoints of this study, was 85% and the lower limit of the 95% confidence interval was 78%, which was above 60% (the percentage pre-determined by objective performance criteria [OPC] minus a non-inferiority margin of 10%), meeting the primary endpoint.

The primary effectiveness endpoint analysis in the ITT population showed that the procedural success rate following treatment with the Pathway PV System alone was 43.5% and the lower limit of the 95% confidence interval was 40.6%, which was below 45% (the percentage pre-determined by 55% of OPC minus a noninferiority margin of 10%), not meeting the primary endpoint. However, the procedural success rate in 116 lesions when the Pathway PV System was used in combination with an adjunctive therapy (PTA or stenting etc.) was 58.8%, which was clinically significant. The procedural success rate in the evaluable subgroup, which was defined as subjects with stenosis diameter ≥ 70% based on an assessment performed in the Angiographic Core Laboratory prior to the procedure, was 50.3%. Although this percentage was below 55% of OPC, the lower limit of the 95% confidence interval was 46.8%, within the range of the non-inferiority margin (45%), indicating that the procedural success rate using Pathway PV System in the subgroup was not inferior to OPC, meeting the primary effectiveness endpoint. In addition, the procedural success rate in 80 lesions when the Pathway PV System was used in combination with an adjunctive therapy (PTA or stenting etc.) was 66.9%. This demonstrated that the Pathway PV System can be used in combination with currently accepted treatment using PTA and stents and be of benefit to patients. The procedural success rate in the ITT population visually assessed by the investigator was 59.7% and the 95% confidence interval was 56.8%— 62.6%, showing significant non-inferiority and superiority to OPC.

The TLR rate using the Pathway PV System in the 6-month post-procedure period was 8.7% (15/172 subjects). No surgical TLRs, deaths, or amputations occurred. No surgical TLRs occurred through 6-month post-procedure. One event of death that was not related to the use of the Pathway PV System and two events of scheduled amputations were reported. No device malfunctions were reported.

The J-SUPREME clinical study was a prospective, multicenter, single arm study conducted using the Jetstream Atherectomy System, in which a total of 60 subjects (50 primary subjects and 10 roll-in subjects) were enrolled at 10 investigational sites in Japan.

The primary endpoint was the primary patency rate at 6 months post index-procedure. Primary vessel patency, a binary endpoint, was defined as follows:

- Bailout stenting or by-pass procedure during the index procedure is not needed (Procedural Success)
- Duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) ≤2.4 at the 6-month follow-up visit, in
  the absence of clinically-driven TLR and/or bypass of the target lesion and/or target limb major
  amputation through 6 months.

Subjects were with symptomatic occlusive atherosclerotic lesions in SFA, PPA and classified as Rutherford category (RC) 2, 3 or 4. Subjects received treatment with the Jetstream Atherectomy System and had stenotic, restenotic or occlusive lesions  $\leq 150$  mm in length and vessel diameter  $\geq 3.0$  mm to  $\leq 6.0$  mm (both by visual estimate). Target lesion had calcified lesions with degree of stenosis  $\geq 70\%$  by visual angiographic assessment or occlusions, regardless of degree of calcification.





### 5. Device Description

The test device is intended to be used to excise and aspirate atherosclerotic disease and hard stenosis from severely calcified lesions (including occlusive lesions) in the SFA and/or PPA.

The Jetstream Atherectomy System is a rotational atherectomy catheter system designed for use in debulking and treating vascular disease in the peripheral vasculature. The catheter includes multiple distal ports located at the catheter tip, which are designed to provide independent infusion and aspiration functions for the active removal of fluid, excised tissue and thrombus from the peripheral treatment site. The Jetstream Atherectomy System consists of two primary components that are packaged separately; Jetstream Atherectomy Catheter set and Jetstream Console (Figure 5-1).



Figure 5-1: Jetstream Atherectomy System

### 5.1. Jetstream Atherectomy Catheter

Jetstream Catheter set is a sterile, single use unit consisting of an electrically driven Catheter and Control Pod with detachable Activation Handle. The Catheter utilizes a differentially cutting tip and includes both aspiration and infusion capabilities. The Activation Handle provides a user interface with keypad controls for device operation. The unit, its electrical connectors, tubing, and aspirant collection bag are packaged in a single pouched tray with retention lid, and sterilized with ethylene oxide (EO). Note that the tray retention lid is not a sterile barrier.

The catheter has four types of model based on existence of expandable blade and size of catheter tip as shown in Table 5-1 and Figure 5-2. The Jetstream single cutter (SC) catheters are available in 1.6 mm and 1.85 mm sizes and the Jetstream expandable cutter (XC) catheters are available in 2.1 mm (Blade Down)/3.0 mm (Blade Up) and 2.4 mm (Blade Down)/3.4 mm (Blade Up). XC model has a mechanism that expandable blade is fold when blade down and expandable blade rises up (i.e. Blade Up) when MAX button in the control pod is turned on.

Table 5-1: Jetstream Specifications

| Model | Tip Diameter | Catheter Length | Minimun Introducer<br>Size | Maximum<br>Guidewire<br>Diameter |
|---|---|---|---|---|
| SC 1.6 | 1.6 mm | 145 cm | 7 Fr | |
| SC 1.85 | 1.85 mm | 145 cm | / [[ | |
| XC 2.1/3.0 | 2.1 mm (Blade Down)<br>3.0 mm (Blade Up) | 135 cm | 7 Fr | 0.014 inch |
| XC 2.4/3.4 | 2.4 mm (Blade Down)<br>3.4 mm (Blade Up) | 120 cm | / [[ | |



Figure 5-2: Jetstream Catheter Tip

#### 5.2. Jetstream Console

A reusable PV Console consists of two (2) peristaltic pumps for aspiration and infusion, power supply, system controller, keypad interface, and LED indicators for device operational status. The PV Console mounts on a standard IV stand and remains outside the sterile field during the procedure (Figure 5-1).

### 5.3. Device Labeling of investigational device

The Directions for Use (DFU) for the Jestream Atherectomy System will be included in the Manual of Operations. The Jetstream catheter and control pod set is labeled on the outer carton. The Jetstream Console is labeled on the product itself. The labeling will include the following information in Japanese or in English.

#### In Japanese:

- Identification number
- Sponsor name and address
- Storage condition
- Exclusively for Clinical Investigations

#### In English:

- Lot number
- Jetstream Catheter model (diameter in mm)
- Expiration (use by) date

### 6. Study Objectives and Endpoints

#### 6.1. Study Objective

The objective of the J-SUPREME II clinical trial is to evaluate the safety and effectiveness of the Boston Scientific (BSC) Jetstream Atherectomy System (Jetstream) for the treatment of Japanese patients with symptomatic occlusive atherosclerotic lesions in native superficial femoral artery (SFA) and/ or proximal popliteal arteries (PPA)

#### 6.2. Primary Endpoint

The primary effective endpoint is the lesion success rate at the index procedure.

Lesion success is defined as the case meets all criteria below:

#### After dilatation with DCB:

- Residual stenosis at the target lesion being ≤30%
- No occurrence of Grade C or greater dissection (NHLBI)

- No occurrence of clinically apparent perforation requiring treatments
- No occurrence of any obstructive complication (e.g., recoil) demonstrating a marked decrease in the flow in the target vessel



### 6.3. Additional Endpoint

Additional endpoints that will be evaluated, but are not necessarily powered to make statistically based conclusions are as follows:

- Procedural success rate (Bailout stenting or by-pass procedure during the index procedure is not needed)
- Rate of distal emboli requiring additional treatment during the procedure or within 24 hours post-index procedure.
- Reduction in lesion stenosis, that is, the difference between the percent stenosis prior to treatment with Jetstream and the percent stenosis following treatment with Jetstream (absolute mean percentage)
- MAE rate at 1 month and 6 months post-index procedure, defined as all-cause death through 1 month, and/or target limb major amputation and/or TLR through 6 months
- Clinically-driven TLR and Target Vessel Revascularization (TVR) Rate at each time point
- Adverse Event rates at each time point
- Distribution of Rutherford Class as compared to baseline at 1 month and 6 months post-index procedure
- Rate of Primary and Secondary Sustained Clinical Improvement as assessed by changes in Rutherford Classification as compared to baseline at 1 month and 6 months post-index procedure
- Rate of Hemodynamic Improvement as assessed by changes in Ankle-Brachial Index as compared to baseline at 1 month and 6 months post-index procedure
- Primary Patency and Assisted Primary Patency at 1 month and 6 months using PSVR 2.4
- Primary Patency and Assisted Primary Patency at 1 month and 6 months using different PSVRs

### 7. Study Design

The J-SUPREME II clinical trial is a prospective, multicenter, single-arm clinical trial of Jetstream Atherectomy System for the treatment of Japanese patients with symptomatic occlusive atherosclerotic lesions in the superficial femoral and/or proximal popliteal arteries.

#### 7.1. Scale and Duration

Thirty-one (31) subjects will be enrolled in the J-SUPREME II clinical trial.

The enrollment period is expected to last approximately 6 months.

The trial will be considered complete (with regards to the primary endpoint) after all enrolled subjects have completed the index procedure, are discontinued prior to completion of the procedure or have died.

The trial will be considered complete (with regards to all follow-up) after all enrolled subjects have completed the 6 month follow-up visit, are discontinued prior to 6 month follow-up visit, have died, or the last 6 month follow-up visit window is closed.

It is estimated that it will take approximately 1 year to complete this trial.



### 7.3. Justification for the Study Design

Pathway PV system which is the first generation model of Jetstream received 510(K) approval in July 2008, and then, the current generation model (Jetstream) in April, 2013. Also, it received CE Mark certification in

September 2013. Jetstream is now commercially available in the U.S., Canada, EU, Australia or other foreign areas except for Japan and its' effectiveness and safety have been confirmed.

J-SUPREME clinical trial was conducted in Japan to evaluate the safety and effectiveness of Jetstream for the treatment of Japanese patients prior to J-SUPREME II clinical trial. Patients with lesions need to be treated with atherectomy device that sufficient revascularization cannot be expected from the PTA alone



### 8. Subject Selection

### 8.1. Study Population and Eligibility

Clinical and angiographic inclusion and exclusion criteria are included in Table8-1 and Table 8-2, respectively. Prior to enrollment, a subject must meet all of the clinical and angiographic inclusion criteria and none of the clinical and angiographic exclusion criteria.

#### 8.2. Inclusion Criteria

Subjects who meet all of the following criteria (see Table 8-1) may be given consideration for inclusion in this clinical investigation, provided no exclusion criterion (see Section 8.3) is met.

Table 8-1: Inclusion Criteria

| Inclusion<br>Criteria | | ≥20 years of age An acceptable candidate for percutaneous intervention and/or emergency surgery. |
|---|---|---|
| | 3. | Willing and able to provide consent before any study specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits |
| | 4. | Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3 or 4 |
| | 5. | Stenotic, restenotic or occlusive lesion(s) located in the native SFA and/or PPA of which meet all of the following criteria*: |





#### 8.3. Exclusion Criteria

Subjects who meet any one of the following criteria (Table 8-2) will be excluded from this clinical study.

Table 8-2: Exclusion Criteria

# Exclusion Criteria

- 1. Target lesion must be one and decided by physician's discretion in the case that eligible lesions exist in both limbs
- 2. Target lesion/vessel with in-stent restenosis
- 3. Target lesion/vessel previously treated with any stent placement prior to the procedure
- 4. Use of atherectomy, laser or other debulking devices other than the Jetstream System, CTO devices or cutting balloon, Angioscore or similar devices, or ultra-high pressure balloon in the target limb SFA/PPA during the index procedure
- 5. History of major amputation in the target limb
- 6. Life expectancy less than 12 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the clinical trial, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the clinical trial
- 7. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated
- 8. Known hypersensitivity/allergy to the investigational atherectomy system or protocol related therapies (e.g., nitinol, stainless steel or other stent materials, and antiplatelet or anticoagulant, thrombolytic medications)

- 9. Subject has a history of coagulopathy or hypercoagulable bleeding disorder
- 10 Subject with untreatable hemorrhagic disease or platelet count <80,000 mm<sup>3</sup> or >600,000 mm<sup>3</sup> as baseline assessment.
- 11. Being on peritoneal dialysis
- 12. History of myocardial infarction, or stroke/cerebrovascular accident (CVA) within 6 months prior to study enrollment
- 13. Unstable angina pectoris at the time of the enrollment
- 14. Pregnancy and/or breast feeding
- 15. Current participation in another investigational drug or device clinical study that has not completed the primary endpoint at the time of enrollment or that clinically interferes with the current study endpoints (Note: studies requiring extended follow-up for products that were investigational, but have become commercially available since then are not considered investigational studies.)
- 16. Septicemia at the time of enrollment
- 17. Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure
- 18. Presence of aneurysm in the target vessel
- 19. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to the index procedure
- 20. Perforated vessel as evidenced by extravasation of contrast media prior to the index procedure



### 9. Subject Accountability

#### 9.1. Point of Enrollment

Once the subject has signed the IRB-approved study ICF, and has met all clinical inclusion and no clinical exclusion criteria, the subject will be considered eligible to be tentatively enrolled in the trial. If the subject is found to meet exclusion criteria during the angiographic eligibility assessment, the subject will be considered a screen failure and should not be enrolled or receive an investigational device, nor should the subject be followed post-procedure per protocol.



### 9.2. Withdrawal

All subjects enrolled in the clinical study (including those withdrawn from the clinical study or lost to follow-up) shall be accounted for and documented.

While trial withdrawal is discouraged, subjects may choose to withdraw from the trial at any time, with or without reason and without prejudice to further treatment. Withdrawn subjects will not undergo any additional trial follow-up, nor will they be replaced (the justified sample size considers an estimated allowance for attrition). The reason for withdrawal will be recorded (if given) in all cases of withdrawal. The Investigator may discontinue a subject from participation in the trial if the Investigator feels that the subject can no longer fully comply with the requirements of the trial or if any of the trial procedures are deemed potentially harmful to the subject. Data that have already been collected on withdrawn subjects will be retained and used for analysis but no new data will be collected after withdrawal.



### 9.4. End-of- Study Definition

The trial will be considered complete (with regards to the primary endpoint) after all enrolled subjects have completed the index procedure, are discontinued prior to completion of the procedure or have died.

The trial will be considered complete (with regards to all follow-up) after all enrolled subjects have completed the 6 month follow-up visit, are discontinued prior to 6 month follow-up visit, have died, or the last 6 month follow-up visit window is closed.

### 10. Study Methods

#### 10.1. Data Collection

The data collection schedule for the J-SUPREME II clinical trial is summarized in Table 10-1.

### 10.2. Study Candidate Screening

A Screening Log will be maintained by each investigational site to document selected information about subjects who fail to meet the J-SUPREME II clinical trial eligibility criteria, including the reason for screen failure.

### 10.2.1. Strategies for Recruitment and Retention

Subjects may be recruited through the investigator's practice, referring physicians and/or the use of recruitment tools. Potential subjects may be identified through an investigational site's database query (chart reviews) or as new or existing patients attend clinic visits. Any information disseminated to potential subjects (eg, advertisements, pamphlets, posters) must be reviewed by the investigational center's IRB/IEC prior to use.

#### 10.3. Informed Consent

Before any study specific tests or procedures are performed, subjects who meet the clinical eligibility criteria will be asked to sign the IRB-approved study ICF. Subjects must be given ample time to review the ICF and have questions answered before signing.

Study personnel should explain to the subject that even if the subject agrees to participate in the trial and signs the ICF, catheterization may demonstrate that the subject is not a suitable candidate for the trial.

Refer to section 9.1 for definition of point of enrollment.





### **Jetstream**

The DFU for the Jetstream Atherectomy System is provided in the Manual of Operations. Prior to use of the device, the treating physician must carefully read and be familiar with the entire DFU. The Jetstream DFU must be followed for performing the device.

Anticoagulant therapy should be consistent with the hospital standard of practice during the procedure.



### 10.13. Follow-up

All enrolled subjects who receive a treatment of Jetstream Atherectomy system will be evaluated prior to discharge from the index procedure and at 1 month and 6 month after the index procedure.





### 11. Statistical Considerations

This section describes statistical approaches of this study. More details will be described in a separate statistical analysis plan.

### 11.1. Endpoints

### 11.1.1. Primary Endpoints

The primary endpoint in this trial is the lesion success rate at the index procedure. Refer to section 6.2 for details.

| The primary endpoint in this | trial is the lesion success rate | at the index procedure. Refer t | o section 6.2 for details |
|---|---|---|---|

| _ |
|---|
| _ |

#### 11.2. General Statistical Methods

### 11.2.1. Analysis Sets

The primary endpoints and additional endpoint / measurements will be analyzed on an Intent- To-Treat (ITT) and a Per-Protocol (PP) basis. All subjects who sign the written informed consent form (ICF) (see Section 19) and are enrolled in the trial (see Section 9.1 for point of enrollment) will be included in the ITT analysis population, regardless of whether the test device is activated. For PP analysis, only subjects who are activated with the test device will be included in the analysis population.

### 11.2.2. Control of Systematic Error/Bias

| All subjects who have met the inclusion/exclusion criteria and signed the | ICF will be eligible for enrollment in |
|---|---|
| the study. | |



### 11.3.4. Justification of Pooling

Not applicable.



### 11.3.6. Other Analyses

Handling of dropouts and missing data will depend on their frequency and the nature of the outcome measure. Sensitivity analyses (e.g., tipping-point analysis) will be performed to assess the impact of subjects with inadequate follow-up (i.e., missing data) on the primary endpoint and to assess the robustness of the conclusion of the primary analysis. Statistical models that account for censored data will be employed in appropriate circumstances (e.g., for time-to-event outcomes). Suspected invalid data will be queried and corrected in the database prior to statistical analysis. Additional information may be found in the Statistical Analysis Plan.

### 11.3.7. Changes to Planned Analyses

Any changes to the planned statistical analyses described above made prior to performing the analyses will be documented in an amended Statistical Analysis Plan approved prior to performing the analyses. Changes from the planned statistical methods after performing the analyses will be documented in the clinical study report along with a reason for the deviation.

#### 12. Data Management

#### 12.1. Data Collection, Processing, and Review

Subject data will be recorded in a limited access secure electronic data capture (EDC) system.

The clinical database will reside on a production server hosted by EDC System. All changes made to the clinical data will be captured in an electronic audit trail and available for review by Boston Scientific Japan K.K. (BSJ) or its representative. The associated RAVE software and database have been designed to meet regulatory compliance for deployment as part of a validated system compliant with laws and regulations applicable to the conduct of clinical studies pertaining to the use of electronic records and signatures. Database backups are performed regularly.

The Investigator provides his/her electronic signature on the appropriate electronic case report forms (eCRFs) in compliance with regulations. Changes to data previously submitted to the sponsor require a new electronic signature by the Investigator acknowledging and approving the changes.

Visual and/or electronic data review will be performed to identify possible data discrepancies. Manual and/or automatic queries will be created in the EDC system and will be issued to the site for appropriate response. Site staff will be responsible for resolving all queries in the database.

#### 12.2. **Data Retention**

The Principal Investigator or his/her desginee and Investigational site will maintain all essential trial documents and source documents, in original format, that support the data collected on study patients in compliance with GCP guidelines. Documents must be retained until the date of the marketing application approval of the test device, or for at least 3 years after the formal discontinuation or completion of the clinical investigation of the device, whichever is longer.

When these documents no longer need to be maintained, it is BSJ's responsibility to inform the Investigator and Site. The Investigator and Site will take measures to ensure that these essential documents are not accidentally damaged or destroyed. If for any reason the Investigator and Site withdraw responsibility for maintaining these essential documents, custody must be transferred to an individual who will assume responsibility. BSJ must receive written notification of this custodial change.

BSJ must maintain necessary essential documents for 5 years from the date of the marketing application approval (or during the period of user-results evaluation, if applicable and if longer than 5 years) or until 3 years have elapsed since the formal discontinuation or completion of the clinical investigation of the device, whichever is longer.



### 13. Deviations

An Investigator must not make any changes or deviate from this protocol, except to protect the life and physical well-being of a subject in an emergency. An investigator shall notify the sponsor and the reviewing IRB of any deviation from the investigational plan to protect the life or physical well-being of a subject in an emergency, and those deviations which affect the scientific integrity of the clinical investigation. Such notice shall be given as soon as possible, but no later than 5 working days after the emergency occurred.

All deviations from the investigational plan, with the reason for the deviation and the date of occurrence, must be documented and reported to the sponsor using EDC. Sites may also be required to report deviations to the IRB, per local guidelines and government regulations.

Deviations will be reviewed and evaluated on an ongoing basis and, as necessary, appropriate corrective and preventive actions (including notification, site re-training, or site discontinuation/termination) will be put into place by the sponsor.

### 14. Device/Equipment Accountability

The investigational devices/equipment shall be securely maintained, controlled, and used only in this clinical study.

BSJ shall keep records to document the physical location of all Jetstream investigational devices from shipment of investigational devices to the investigation sites until return or disposal.

The principal investigator or an authorized designee shall keep records documenting the receipt, use, return and disposal of the Jetstream investigational devices, which shall include the following:

- Date of receipt
- Identification of each investigational device (Lot number or unique code)
- Expiry date, as applicable
- Date or dates of use
- Subject identification
- Date on which the investigational device was returned, if applicable
- Date of return (and number) of unused, expired, or malfunctioning investigational devices, if applicable.
- Date on which the investigational device was discarded, if applicable

Once the Investigator and Site are notified by BSJ that subject enrollment is complete, all unused test devices and/or accessories must be returned to BSJ.

### 15. Compliance

### 15.1. Statement of Compliance

The J-SUPREME II clinical trial will be conducted in accordance with the ethical principles that have their origins in the Declaration of Helsinki and that are consistent with Good Clinical Practices (GCP), Order for Enforcement of the Pharmaceutical and Medical Device Law, regulatory requirements and this protocol. The study shall not begin until the required approval from the IRB and/or favorable opinion from regulatory authority has been obtained, if appropriate. Also, the study shall not begin prior to issuance of the site Authorization to Enroll, as provided by BSJ. Any additional requirements imposed by the IRB or regulatory authority shall be followed, if appropriate.

### 15.2. Investigator Responsibilities

The Principal Investigator of an investigational site is responsible for ensuring that the study is conducted in accordance with the Clinical Study Agreement, the clinical investigational plan, GCP, ethical principles that have their origins in the Declaration of Helsinki, any conditions of approval imposed by the reviewing IRB, and Pharmaceutical and Medical Device Act, Regulatory authority, whichever affords the greater protection to the subject.

The Principal Investigator's responsibilities include, but are not limited to, the following.

- Prior to beginning the study, confirm the Clinical Study Agreement and comply with the Investigator responsibilities as described in such Agreement.
- Prior to beginning the study, sign protocol signature page documenting his/her agreement to conduct the study in accordance with the protocol.
- Provide his/her qualifications and experience to assume responsibility for the proper conduct of the study
  and that of key members of the site team through up-to-date curriculum vitae or other relevant
  documentation.
- Make no changes in or deviate from this protocol, except to protect the life and physical well-being of a subject in an emergency; document and explain any deviation from the approved protocol that occurred during the course of the clinical investigation.

- Create and maintain source documents throughout the clinical study and ensure their availability with direct
  access during monitoring visits or audits; ensure that all clinical-investigation-related records are retained
  per requirements.
- Ensure the accuracy, completeness, legibility, and timeliness of the data reported to the sponsor in the CRFs and in all required reports.
- Record, report, and assess (seriousness and relationship to the device/procedure) every adverse event as applicable per the protocol and observed device deficiency.
- Report to sponsor, per the protocol requirements, all SAEs and device deficiencies that could have led to a SADE and potential/USADE.
- Report to the IRB any SAEs and device deficiencies that could have led to a SADE and potential/USADE,
  if required by applicable laws or regulations or this protocol or by the IRB, and supply BSJ with any
  additional requested information related to the safety reporting of a particular event.
- Maintain the device accountability records and control of the device, ensuring that the investigational device
  is used only by authorized/designated users and in accordance with this protocol and instructions/directions
  for use.
- Allow the sponsor to perform monitoring and auditing activities, and be accessible to the clinical research monitor or auditor and respond to questions during monitoring visits or audit(s).
- Allow and support regulatory authorities and the IRB when performing auditing activities.
- Ensure that informed consent is obtained in accordance with applicable laws, this protocol and local IRB requirements.
- Provide adequate medical care to a subject during and after a subject's participation in a clinical study in the case of adverse events, as described in the Informed Consent Form (ICF).
- Inform the subject of the nature and possible cause of any adverse events experienced.
- Inform the subject of any new significant findings occurring during the clinical investigation, including the need for additional medical care that may be required.
- Ensure that clinical medical records are clearly marked to indicate that the subject is enrolled in this clinical study.
- Ensure that, if appropriate, subjects enrolled in the clinical investigation are provided with some means of showing their participation in the clinical investigation, together with identification and compliance information for concomitant treatment measures (contact address and telephone numbers shall be provided).
- Inform, with the subject's approval or when required by national regulations, the subject's personal physician about the subject's participation in the clinical investigation.
- Make all reasonable efforts to ascertain the reason(s) for a subject's premature withdrawal from clinical investigation while fully respecting the subject's rights.
- Ensure that an adequate investigational site team and facilities exist and are maintained and documented during the clinical investigation.

#### 15.2.1. Delegation of Responsibility

When specific tasks are delegated by an investigator, including but not limited to conducting the informed consent process, the Principal Investigator is responsible for providing appropriate training, are competent to perform the tasks they have been delegated and adequate supervision of those to whom tasks are delegated. Where there is a sub investigator at a site, the sub investigator should not be delegated the primary supervisory responsibility for the site. The investigator is accountable for regulatory violations resulting from failure to adequately supervise the conduct of the clinical study.

#### 15.3. Institutional Review Board

The investigational site will obtain the written and dated approval/favorable opinion of the IRB for the clinical investigation before recruiting subjects and implementing all subsequent amendments, if required.

Page 36 of 56

The written IRB approval of the protocol and Informed Consent Form, must be received by the sponsor before recruitment of subjects into the study and shipment of investigational products/equipment. Prior approval must also be obtained for other materials related to subject recruitment or which will be provided to the subject.

Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All changes to the ICF will be IRB approved; a determination will be made regarding whether a new ICF needs to be obtained from participants who provided consent, using a previously approved ICF. Annual IRB approval and renewals will be obtained throughout the duration of the study as required by IRB requirements. Copies of the Investigator's reports and/or the IRB continuance of approval must be provided to the Sponsor.

### 15.4. Sponsor Responsibilities

The clinical trial organization in Japan, including investigational sites in Japan, is provided as an attachment to the protocol.

All information and data sent to BSJ and its authorized designee concerning subjects or their participation in this study will be considered confidential by BSJ and will be kept confidential in accordance with all applicable laws and regulations. Only authorized BSJ personnel, and/or a BSJ representative including, but not limited to Contract Research Organization (CRO), will have access to this information. Authorized regulatory personnel have the right to inspect and copy all records pertinent to this study. Study data collected during this study may be used by BSJ for the purposes of this study, publication, and to support future research and/or other business purposes, such as overseeing and improving the performance of its device, new medical research and proposals for developing new medical products and procedures. All data used in the analysis and reporting of this study or shared with a third-party researcher will be without identifiable reference to specific subjects.

Information received during the study will not be used to market to subjects; subject names will not be placed on any mailing lists or sold to anyone for marketing purposes.

**Note:** BSJ may utilize a contract research organization (CRO) or other contractors to act as its representative for carrying out designated tasks. Responsibilities for these entities are defined in the applicable contracts or agreements. Contact information for the CROs is provided as an attachment to the protocol or in the study Manual of Operations (MOP).



### 15.5. Reimbursement and Compensation

Subject Reimbursement: Travel and other expenses incurred by subjects as a result of participation in the study will be reimbursed in accordance with pertinent Regulations and per the investigational sites.

Compensation for Subject's Health Injury: BSJ will stipulate an insurance policy to cover potential health injury for study subjects. If any study related health injury occurs and a site is held responsible for its compensation, BSJ will assume the responsibility, except in the case those damages are incurred due to intentional misconduct or negligence at the site.
## 16. Monitoring

Monitoring will be performed during the study according to the monitoring plan to assess continued compliance with the protocol and applicable regulations. In addition, the clinical research monitor verifies that study records are adequately maintained, that data are reported in a satisfactory manner with respect to timeliness, adequacy, and accuracy, and that the Principal Investigator continues to have sufficient staff and facilities to conduct the study safely and effectively.

The Investigator/institution guarantees direct access to original source documents by BSJ personnel, CRO or other contractors, and appropriate regulatory authorities. In the event that the original medical records cannot be obtained for a subject that is seen by a non-study physician at a non-study institution, all reasonable attempts must be made to obtain photocopies of the original source documents for review. Photocopies of original source documents related to IMR events that are adjudicated by the IMR (from either the study site or a non-study institution, if applicable) must also be made available for submission to the sponsor Safety Group.

The study may also be subject to a quality assurance audit by BSJ, CRO or other contractors, as well as inspection by appropriate regulatory authorities. It is important that the Investigator and relevant study personnel are available during on-site monitoring visits or audits and that sufficient time is devoted to the process.





#### 17.2. Risks associated with Participation in the Clinical Study

There may be additional risks linked to the procedure, and follow-up testing which are unforeseen at this time. All testing planned for the follow-up period is standard of care.



#### 17.4. Risk Minimization Actions

Additional risks may exist. Risks can be minimized through compliance with this protocol, performing procedures in the appropriate hospital environment, adherence to subject selection criteria, close monitoring of the subject's physiologic status during research procedures and/or follow-ups and by promptly supplying BSJ with all pertinent information required by this protocol.

#### 17.5. Anticipated Benefits

Potential anticipated benefits include the improvement of procedural success of atherosclerotic SFA/PPA lesions with improvement in the symptoms of disease. However, the Jetstream Atherectomy system is an investigational device and these potential benefits may or may not actually be present.

## 17.6. Risk to Benefit Rationale

The Jetstream system is expected to be suitable for its intended purpose. There are no unacceptable residual risks/intolerable risks and all applicable risks have been addressed through the provision of appropriate Directions for Use (DFU) and Kiki-Gaiyosho. Evaluation of the risks and benefits that are expected to be associated with the use of the Jetstream Atherectomy system demonstrate that when used under the conditions intended, the benefits associated with the use of the Jetstream Atherectomy system should outweigh the risks in Japan.

## 18. Safety Reporting

## 18.1. Reportable Events by investigational site to Boston Scientific

It is the responsibility of the investigator to assess and report to BSJ any event which occurs in any of following categories:

- All Serious Adverse Events (SAE)
- All Investigational Device Deficiencies
- Unanticipated Serious Adverse Device Effects (USADE)/ Unanticipated Adverse Device Effects (UADE)
- Adverse Device Effect (ADE)/ Serious Adverse Device Effect (SADE)
- New findings/updates in relation to already reported events













#### 18.5. Boston Scientific Device Deficiencies

All investigational device deficiencies (including but not limited to failures, malfunctions, use errors, product nonconformities, and inadequacy in the information supplied by the manufacturer) regarding Jetstream Atherectomy System will be documented and reported to BSC. If possible, the device(s) should be returned to BSC for analysis. Instructions for returning the investigational device(s) will be provided in the Manual of Operations. If it is not possible to return the device, the investigator should document why the device was not returned and the final disposition of the device. Device failures and malfunctions should also be documented in the subject's medical record.

Device deficiencies (including but not limited to failures, malfunctions, and product nonconformities) are not to be reported as adverse events. However, if there is an adverse event that results from a device failure or malfunction, would be recorded as an adverse event on the appropriate eCRF.

Any Investigational Device Deficiency that might have led to a SAE if a) suitable action had not been taken or b) intervention had not been made or c) if circumstances had been less fortunate is considered a reportable event.

#### 18.6. Reporting to Regulatory Authorities / IRBs / Investigators

BSJ will report to regulatory agency and notify all PIs and head of the investigational sites if any significant safety information was received. Additionally, information which implies possible influence to patient's safety and the conduct of the study will also notified to all PIs and the head of the investigational sites.

## 19. Informed Consent

Subject participation in this clinical study is voluntary. Informed Consent is required from each subject. The Investigator is responsible for ensuring that Informed Consent is obtained prior to the use of any investigational devices, study-required procedures and/or testing, or data collection.

The obtaining and documentation of Informed Consent must be in accordance with the ethical principles that have their origins in the Declaration of Helsinki and that are consistent with Good Clinical Practices (GCP), Pharmaceutical Affairs Law, regulatory authority and this protocol. The ICF must be accepted by BSJ or its delegate (e.g. CRO), and approved by the site's IRB, or central IRB, if applicable.

Boston Scientific Japan K.K. will provide a study-specific template of the ICF to investigators participating in this study. The ICF template may be modified to meet the requirements of the investigative site's IRB. Any modification requires acceptance from BSJ prior to use of the form. The ICF must be in a language understandable to the subject and if needed. Privacy language shall be included in the body of the form or as a separate form as applicable.

The process of obtaining Informed Consent shall at a minimum include the following steps, as well as any other steps required by applicable laws, rules, regulations and guidelines:

- be conducted by the Principal Investigator or designee authorized to conduct the process,
- include a description of all aspects of the clinical study that are relevant to the subject's decision to participate throughout the clinical study,
- avoid any coercion of or undue influence of subjects to participate,
- not waive or appear to waive subject's legal rights,
- use native language that is non-technical and understandable to the subject,
- provide ample time for the subject to consider participation and ask questions if necessary,
- ensure important new information is provided to new and existing subjects throughout the clinical study.

The ICF shall always be signed and personally dated by the subject to sign the ICF under the applicable laws, rules, regulations and guidelines and by the investigator and/or an authorized designee responsible for conducting the informed consent process. If a legal representative signs, the subject shall be asked to provide informed consent for continued participation as soon as his/her medical condition allows. The original signed ICF will be retained by the site and a copy of the signed and dated document and any other written information must be given to the person signing the form. Informed Consent signature can be replaced by printed name and seals of appropriate individuals.

If new information becomes available that can significantly affect a subject's future health and medical care, that information shall be provided to the affected subject(s) in written form via a revised ICF or, in some situations, enrolled subjects may be requested to sign and date an addendum to the ICF. In addition to new significant information during the course of a study, other situations may necessitate revision of the ICF, such as if there are amendments to the applicable laws, protocol, a change in Principal Investigator, administrative changes, or following annual review by the IRB. The new version of the ICF must be approved by the IRB. Acceptance by Boston Scientific Japan K.K. is required if changes to the revised ICF are requested by the site's IRB. The IRB will determine the subject population to be re-consented.

Study personnel should explain to the subject that even if the subject agrees to participate in the trial and signs the ICF, catheterization may demonstrate that the subject is not a suitable candidate for the trial. A Screening Log will be maintained by the investigational site to document select information about candidates who fail to meet the trial eligibility criteria, including, but not limited to, the reason for screen failure.

## 20. Committees

#### 20.1. Executive Committee

An Executive Committee composed of BSC/BSJ Clinical Management and selected Coordinating Principal Investigator(s) will be convened. This committee will be responsible for the overall conduct of the study which will include protocol development, study progress, subject safety, overall data quality and integrity, and timely dissemination of study results through appropriate scientific sessions and publications. As appropriate the Executive Committee may request participation of J-SUPREME II clinical trial Investigators on the committee.



## 21. Suspension or Termination

## 21.1. Premature Termination of the Study

Boston Scientific Japan K.K. reserves the right to discontinue or terminate the study at any stage but intends to exercise this right only for valid scientific or administrative reasons and reasons related to protection of subjects. Investigators, associated IRBs, and regulatory authorities, as applicable, will be notified in writing in the event of study termination or discontinuation.

#### 21.1.1. Criteria for Premature Termination of the Study

Possible reasons for study discontinuation or termination include, but are not limited to, the following.

- The occurrence of unanticipated adverse device effects that present a significant or unreasonable risk to subjects enrolled in the study.
- An enrollment rate far below expectation that prejudices the conclusion of the study.
- A decision on the part of Boston Scientific Japan K.K. to suspend or discontinue development of the device.

# 21.2. Termination of Study Participation by the Investigator or Withdrawal of IRB Approval

Any investigator or IRBs in the J-SUPREME II clinical trial may discontinue participation in the study or withdrawal approval of the study, respectively, with suitable written notice to BSJ. Investigators, associated IRBs, and regulatory authorities, as applicable, will be notified in writing in the event of these occurrences.

### 21.3. Requirements for Documentation and Subject Follow-up

In the event of premature study termination a written statement as to why the premature termination has occurred will be provided to all participating sites by BSJ. The IRB and regulatory authorities, as applicable, will be notified. Detailed information on how enrolled subjects will be managed thereafter will be provided.

In the event an IRB terminates participation in the study, participating investigators, associated IRBs, and regulatory authorities, as applicable, will be notified in writing. Detailed information on how enrolled subjects will be managed thereafter will be provided by BSJ.

In the event a Principal Investigator terminates participation in the study, study responsibility will be transferred to another investigator, if possible. In the event there are no opportunities to transfer Principal Investigator responsibility; detailed information on how enrolled subjects will be managed thereafter will be provided by BSJ.

Also, the Principal Investigator or his/her designee must return all study-related documents and investigational product to Boston Scientific, unless this action would jeopardize the rights, safety, or welfare of the subjects.

#### 21.4. Criteria for Suspending/Terminating a Study Site

BSJ reserves the right to stop the inclusion of subjects at investigational site at any time after the study initiation visit if no subjects have been enrolled for a period beyond 3 months after site initiation, or if the site has multiple or severe protocol violations/noncompliance without justification and/or fails to follow remedial actions.

In the event of termination of site participation, all study devices and testing equipment, as applicable, will be returned to BSJ unless this action would jeopardize the rights, safety or well-being of the subjects. The IRB and regulatory authorities, as applicable, will be notified. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

## 22. Publication Policy

BSJ requires disclosure of its involvement as a sponsor or financial supporter in any publication or presentation relating to a BSJ study or its results. BSJ will submit study results for publication (regardless of study outcome) in a timely manner. Boston Scientific Corporation follows authorship principals as set forth in the Uniform Requirements of the International Committee of Medical Journal Editors (ICMJE; <a href="http://www.icmje.org">http://www.icmje.org</a>). In order to ensure the public disclosure of study results in a timely manner, while maintaining an unbiased presentation of study outcomes, BSC personnel may assist authors and investigators in publication preparation provided the following guidelines are followed.

- All authorship and contributorship requirements as described above must be followed.
- BSJ involvement in the publication preparation and the BSC Publication Policy should be discussed with the Coordinating Principal Investigator(s) at the onset of the project.
- The First and Senior authors are the primary drivers of decisions regarding publication content, review, approval, and submission.



## 24. Abbreviations and Definitions

## 24.1. Abbreviations

Abbreviations are shown in Table 24-1.

Table 24-1: Abbreviations

| Abbreviation | Terminology |
|--------------|-----------------------------------------------------|
| ABI | Ankle Brachial Index |
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| BSC | Boston Scientific Corporation |
| BSJ | Boston Scientific Japan K.K. |
| CE | Conformité Européenne (meaning European Conformity) |
| CIN | Contrast-Induced Nephropathy |
| CRA | Clinical Research Associate |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CVA | Cerebrovascular Accident |
| DFU | Directions for Use |
| DUS | Duplex Ultrasound |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| eGFR | Estimated Glemerular Filtration Rate |
| EVT | Endovascular Therapy |
| GCP | Good Clinical Practice |
| НСР | Health Care Professional |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IMR | Independent Medical Reviewer |
| ITT | Intent to Treat |
| IRB | Institutional Review Board |
| IVUS | Intravascular Ultrasound |
| MAE | Major Adverse Event |
| OPC | Objective Performance Criteria |
| PAD | Peripheral arterial disease |
| PG | Performance Goal |
| PMDA | Pharmaceutical Medical Device Agency |
| PPA | Proximal Popliteal Artery |

| Abbreviation | Terminology |
|--------------|---------------------------------------------|
| PSVR | Peak Systolic Velocity Ratio |
| PTA | Percutaneous Transluminal Angioplasty |
| QA | Quantitative Angiography |
| QOL | Quality of Life |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SC | Single Cutter |
| SFA | Superficial Femoral Artery |
| TASC | Transatlantic Inter-Societal Concensus |
| TBI | Toe Brachial Index |
| TLR | Target Lesion Revascularization |
| TVR | Target Vessel Revascularization |
| USADE | Unanticipated Serious Adverse Device Effect |
| UPN | Universal Product Number |
| XC | Expandable Cutter |





| I - |
|-----|
| 1 |



